CLINICAL TRIAL: NCT07018986
Title: The MIND-BC Study: MIND Diet for Breast Cancer Cognition
Acronym: MIND-BC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-23571; R01CA299480 (NIH)
Record Dates: First submitted 2025-05-28; First posted 2025-06-13 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MIND Diet Arm (Experimental): Participants (N=200) will be randomized 1:1 to a 12-week intervention phase. The MIND diet arm will be asked to participate in weekly "check-in" sessions with a diet coach supervised by a registered dietitian. To evaluate the longer-term effects of the MIND diet as a part of lifestyle change, we will also conduct a 3-month follow-up assessment.
  Interventions: Other: MIND Diet
- Usual Diet Arm (Active Comparator): Participants (N=200) will be randomized 1:1 to a 12-week intervention phase. The usual diet participants will be provided with weekly grocery gift cards to purchase foods that follow their "usual" diet. Usual diet participants will also conduct a 3-month follow-up assessment.
  Interventions: Other: Usual Diet

INTERVENTIONS:
Other: MIND Diet — a combination of the Mediterranean and DASH diets emphasizing consumption of high-nutrient, plant-based foods such as green leafy vegetables, nuts, berries, fish, and olive oil while limiting intake of foods high in saturated fat, pre-processed snacks, sugar, red and processed meat.
  Other Names: The "Mediterranean-DASH Intervention for Neurodegenerative Delay" (MIND) diet
  Arms: MIND Diet Arm
Other: Usual Diet — Check-in sessions for the usual diet arm will focus on general health (e.g., healthy hair, skin, eyesight). None of the topics will include dietary information for the usual diet arm.
  Arms: Usual Diet Arm

SUMMARY:
This fully, powered efficacy RCT, the MIND diet for Breast Cancer Cognition (MIND-BC), will evaluate the MIND diet in a rigorous, highly controlled academic cancer center. We will recruit breast cancer survivors reporting CRCI with a MIND diet score < 8, based on a previously devised 14-item diet questionnaire designed to detect inadequate diet with respect to brain health (scores range from 0 to 14, with lower scores indicating a less adequate diet).14 Breast cancer survivors will have recently completed adjuvant treatment (i.e., 6 months to three years previously), to ensure that perceived cognitive impairment is likely chronic and due to cancer. To achieve maximal effect, the study consists of two 12-week phases 1) intervention phase, 2) maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with stage I-III breast cancer.
* Able to speak and read English.
* Able to consume foods orally.
* >18 years of age.
* Able to provide informed consent.
* Have no documented or observable psychiatric or neurological disorder that would interfere with study participation (e.g., schizophrenia).
* Report 'somewhat' to 'very much' cognitive impairment in the past week (i.e., a score ≥ 2 on a 0-4 scale) that they attribute to cancer or its treatment.
* Report a MIND diet score < 10 (range 0 to 14, higher score equates to higher diet quality).
* Willing to consume the MIND diet.
* Completed adjuvant treatment 6 months to three years previously.

Exclusion Criteria:

* Not meeting all of the inclusion criteria.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of the MIND diet: Self-reported cognition | At 12 weeks and 3 months
  The Functional Assessment of Cancer Therapy - General (FACT-G) will be used to determine self-reported cognition.

SECONDARY OUTCOMES:
Efficacy of the MIND diet: Fatigue | At 12 weeks and 3 months
  The Functional Assessment of Chronic Illness Fatigue Subscale (FACIT Fatigue) will be used to determine fatigue.
Efficacy of the MIND diet: Quality of life (QOL) and mood | At 12 weeks and 3 months
  The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life of Cancer Patients Questionnaire will be used to determine QOL and mood.
Efficacy of the MIND diet: Objective cognition | At Baseline, 12 weeks, and 3 months
  Neuropsychological tests (i.e., best objective performance) will be administered via the CANTAB Connect (Cambridge Cognition, Cambridge, UK) that contains a well-validated battery of tests based in neuropsychology and neuroscience administered in a semi-automated manner via the web that is automatically scored upon completion. EMA Participants will complete 3 prompted surveys and sets of EMA cognitive tasks throughout the day as well as an end of day survey each day for 7 days at baseline, 12 weeks, and 3 month follow-up including symbol search, dot memory test, shopping list associate test. All scores will be correlated to determine objective cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Crowder, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States